CLINICAL TRIAL: NCT04767529
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Efruxifermin in Non-Cirrhotic Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Study of Efruxifermin in Non-Cirrhotic Subjects With Histologically Confirmed Nonalcoholic Steatohepatitis (NASH)
Acronym: Harmony
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akero Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK-US-001-0102
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- placebo (Placebo Comparator): double-blind, once-weekly subcutaneous injection
  Interventions: Drug: Placebo
- Efruxifermin 28 mg (Experimental): double-blind, once-weekly subcutaneous injection
  Interventions: Drug: Efruxifermin
- Efruxifermin 50 mg (Placebo Comparator): double-blind, once-weekly subcutaneous injection
  Interventions: Drug: Efruxifermin

INTERVENTIONS:
Drug: Efruxifermin — subcutaneous injection
  Other Names: EFX
  Arms: Efruxifermin 28 mg; Efruxifermin 50 mg
Drug: Placebo — subcutaneous injection
  Arms: placebo

SUMMARY:
This is a multi-center evaluation of efruxifermin (EFX) in a randomized, double-blind, placebo-controlled study in non-cirrhotic subjects with biopsy-proven F2 - F3 NASH.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females between 18 - 75 years of age inclusive, based on the date of the screening visit.
* Previous history or presence of 2 out of 4 components of metabolic syndrome (obesity, dyslipidemia, elevated blood pressure, elevated fasting glucose) or type 2 diabetes.
* FibroScan measurement > 8.5 kPa [kilopascal].
* Biopsy-proven NASH. Must have had a liver biopsy obtained ≤ 180 days prior to randomization with fibrosis stage 2 to 3 and a non-alcoholic fatty liver disease (NAFLD) activity score (NAS) of ≥ 4 with at least a score of 1 in each of the following NAS components:

  * Steatosis (scored 0 to 3),
  * Ballooning degeneration (scored 0 to 2), and
  * Lobular inflammation (scored 0 to 3).

Exclusion Criteria:

* Weight loss > 5% in the 3 months prior to screening until randomization or from the time of the diagnostic liver biopsy until randomization, whichever is longer.
* Presence of cirrhosis on liver biopsy (stage 4 fibrosis).
* Type 1 or uncontrolled Type 2 diabetes.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akero Study Director, Study Director — Study Director
Locations (48):
- United States (47):
  - Akero Clinical Study Site, Chandler, Arizona
  - Akero Clinical Study Site, Glendale, Arizona
  - Akero Clinical Study Site, Tucson, Arizona
  - Akero Clinical Study Site, North Little Rock, Arkansas
  - Akero Clinical Study Site, Chula Vista, California
  - Akero Clinical Study Site, Fresno, California
  - Akero Clinical Study Site, La Jolla, California
  - Akero Clinical Study Site, Los Angeles, California
  - Akero Clinical Study Site, Orange, California
  - Akero Clinical Study Site, Panorama City, California
  - Akero Clinical Study Site, Rialto, California
  - Akero Clinical Study Site, Santa Ana, California
  - Akero Clinical Study Site, Fort Myers, Florida
  - Akero Clinical Study Site, Inverness, Florida
  - Akero Clinical Study Site, Lakewood Rch, Florida
  - Akero Clinical Study Site, Miami, Florida
  - Akero Clinical Study Site, Miami Lakes, Florida
  - Akero Clinical Study Site, Ocala, Florida
  - Akero Clinical Study Site, Sarasota, Florida
  - Akero Clinical Study Site, Marietta, Georgia
  - Akero Clinical Study Site, Topeka, Kansas
  - Akero Clinical Study Site, Baton Rouge, Louisiana
  - Akero Clinical Study Site, Marrero, Louisiana
  - Akero Clinical Study Site, Ypsilanti, Michigan
  - Akero Clinical Study Site, Flowood, Mississippi
  - Akero Clinical Study Site, Jackson, Mississippi
  - Akero Clinical Study Site, Las Vegas, Nevada
  - Akero Clinical Study Site, Charlotte, North Carolina
  - Akero Clinical Study Site, Durham, North Carolina
  - Akero Clinical Study Site, Morehead City, North Carolina
  - Akero Clinical Study Site, Cincinnati, Ohio
  - Akero Clinical Study Site, Greenville, South Carolina
  - Akero Clinical Study Site, Hermitage, Tennessee
  - Akero Clinical Study Site, Nashville, Tennessee
  - Akero Clinical Study Site, Arlington, Texas
  - Akero Clinical Study Site, Austin, Texas
  - Akero Clinical Study Site, Cedar Park, Texas
  - Akero Clinical Study Site, Dallas, Texas
  - Akero Clinical Study Site, Edinburg, Texas
  - Akero Clinical Study Site, Fort Worth, Texas
  - Akero Clinical Study Site, Garland, Texas
  - Akero Clinical Study Site, Houston, Texas
  - Akero Clinical Study Site, San Antonio, Texas
  - Akero Clinical Study Site, San Marcos, Texas
  - Akero Clinical Study Site, Webster, Texas
  - Akero Clinical Study Site, Charlottesville, Virginia
  - Akero Clinical Study Site, Richmond, Virginia
- Akero Clinical Study Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrison SA, Frias JP, Neff G, Abrams GA, Lucas KJ, Sanchez W, Gogia S, Sheikh MY, Behling C, Bedossa P, Shao L, Chan D, Fong E, de Temple B, Shringarpure R, Tillman EJ, Rolph T, Cheng A, Yale K; HARMONY Study Group. Safety and efficacy of once-weekly efruxifermin versus placebo in non-alcoholic steatohepatitis (HARMONY): a multicentre, randomised, double-blind, placebo-controlled, phase 2b trial. Lancet Gastroenterol Hepatol. 2023 Dec;8(12):1080-1093. doi: 10.1016/S2468-1253(23)00272-8. Epub 2023 Oct 3. PMID 37802088
- [Derived] Noureddin M, Frias JP, Neff GW, Lucas KJ, Behling C, Bedossa P, Dubourg J, Chan D, Burch M, Fong E, de Temple B, Minerva M, Barrett K, Shringarpure R, Tillman EJ, Rolph T, Cheng A, Yale K. Safety and efficacy of once-weekly efruxifermin versus placebo in metabolic dysfunction-associated steatohepatitis (HARMONY): 96-week results from a multicentre, randomised, double-blind, placebo-controlled, phase 2b trial. Lancet. 2025 Aug 16;406(10504):719-730. doi: 10.1016/S0140-6736(25)01073-6. PMID 40818852

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo; Efruxifermin 28 mg; Efruxifermin 50 mg: double-blind, once-weekly subcutaneous administration
Period: Overall Study
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Started (Randomized (randomly assigned to groups)) | 43 | 42 | 43
Started Study Drug (received at least 1 dose) | 43 | 40 | 43
Completed Week 96 Treatment | 34 | 26 | 27
Discontinued Treatment (Subjects that were randomized but not dosed were included under required use of a prohibited concomitant medication and lost to follow-up for primary reason for discontinuation of treatment) | 9 | 16 | 16
Completed Week 24 Visit | 42 | 37 | 36
Completed (Completed the study) | 34 | 27 | 27
Not Completed | 9 | 15 | 16
Not completed — Adverse Event | 0 | 4 | 3
Not completed — clinical outcomes endpoint (excluding death) | 1 | 3 | 3
Not completed — Required use of a prohibited medication | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 5 | 4
Not completed — At the discretion of the Investigator or Sponsor for noncompliance | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Randomly assigned to groups
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg | Total
Number analyzed (Participants) | 43 | 42 | 43 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 31 | 37 | 102
  >=65 years | 9 | 11 | 6 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (10.1) | 56.5 (9.3) | 52.4 (11.4) | 54.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 23 | 79
  Male | 16 | 13 | 20 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 17 | 20 | 52
  Not Hispanic or Latino | 28 | 25 | 23 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 39 | 38 | 41 | 118
  Race: Black or African American | 2 | 1 | 1 | 4
  Race: Asian | 2 | 3 | 0 | 5
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: American Indian or Alaskan Native | 0 | 0 | 0 | 0
  Race: Other | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 43 | 42 | 43 | 128
Baseline Fibrosis Stage [Count of Participants; unit: Participants] — NASH CRN fibrosis score (scored by a fibrosis score of 0-4, where 0 = no fibrosis, 1 = centrilobular pericellular fibrosis, 2 = centrilobular and periportal fibrosis, 3 = bridging fibrosis, 4 = cirrhosis)
  Participants
    Fibrosis stage 2 | 13 | 15 | 16 | 44
    Fibrosis stage 3 | 30 | 27 | 27 | 84
Weight [Mean (Standard Deviation); unit: kg] — Population: Baseline weight not available for 2 participants
  kg
    number analyzed (Participants) | 43 | 40 | 43 | 126
    (all) | 107.6 (25.6) | 103.9 (22.7) | 102.8 (21.1) | 104.8 (23.2)
Type 2 diabetes status [Count of Participants; unit: Participants]
  T2D yes | 28 | 32 | 30 | 90
  T2D no | 15 | 10 | 13 | 38

OUTCOME MEASURES:

1. Primary Outcome: Effect of Efruxifermin (EFX) vs Placebo on Fibrosis Regression in Participants With Metabolic Dysfunction-associated Steatohepatitis (MASH)-Associated Stage 2 or 3 Fibrosis (F2 or F3)
Description: Proportions of subjects in EFX vs placebo groups with improvement in liver fibrosis, defined as ≥ 1 stage NASH Clinical Research Network [CRN] fibrosis score (score ranges from 0 to 4, increasing with fibrosis severity), and no worsening of steatohepatitis (no increase in NASH Activity Score [NAS], which ranges from 0 to 8 and is the sum of scores of steatosis, lobular inflammation, and hepatocyte ballooning), at Week 24
Time Frame: 24 Weeks
Population: Week 24 Liver Biopsy Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 41 | 38 | 34
Participants | 8 | 15 | 14
Statistical Analysis 1: Comparison: Placebo vs Efruxifermin 28 mg; Comparison between proportion of participants in efruxifermin 28 mg group who met the primary endpoint vs the placebo group; Test type: Superiority; p = 0.025, Cochran-Mantel-Haenszel — Threshold for significance set at p<0.05; Cochran-Mantel-Haenszel test adjusting for stratification factors was used for comparison between the EFX 28 mg and placebo group; percent difference = 22.6, 95% CI 2-sided [3.8 to 41.4] — % difference from placebo (efruxifermin 28 mg - placebo)
Statistical Analysis 2: Comparison: Placebo vs Efruxifermin 50 mg; Comparison between proportion of participants in efruxifermin 50 mg group who met the primary endpoint vs the placebo group; Test type: Superiority; p = 0.036, Cochran-Mantel-Haenszel — Threshold for significance was p<0.05; Cochran-Mantel-Haenszel test adjusting for stratification factors is used for comparison between the EFX 50 mg and placebo group; percent difference = 22.5, 95% CI 2-sided [1.6 to 43.3] — % difference from placebo (efruxifermin 50 mg - placebo)

2. Secondary Outcome: Proportion of Subjects Who Achieve Improvement in Liver Fibrosis ≥ 1 Stage and no Worsening of Steatohepatitis at Week 96
Description: Proportions of subjects in EFX vs baseline groups who achieve improvement in liver fibrosis (decrease of ≥ 1 stage in NASH CRN fibrosis score) and no worsening of steatohepatitis (no increase in NAS for ballooning, inflammation, or steatosis) at Week 96
Time Frame: 96 Weeks
Population: Week 96 Liver Biopsy Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 34 | 26 | 28
Participants | 8 | 12 | 21
Statistical Analysis 1: Comparison: Placebo vs Efruxifermin 28 mg; Test type: Superiority; p = 0.070, Cochran-Mantel-Haenszel — Threshold for significance set at p<0.05; A Cochran-Mantel-Haenszel test adjusting for stratification factors was used for comparisons between the efruxifermin 28 mg and placebo group; percent difference = 21.8, 95% CI 2-sided [-1.3 to 45.0]
Statistical Analysis 2: Comparison: Placebo vs Efruxifermin 50 mg; Week 96; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Threshold for significance set at p<0.05; A Cochran-Mantel-Haenszel test adjusting for stratification factors was used for comparisons between the efruxifermin 50 mg and placebo group; percent difference = 51.9, 95% CI 2-sided [31.2 to 72.7]

3. Secondary Outcome: Proportion of Subjects Who Achieve Resolution of Steatohepatitis and no Worsening of Liver Fibrosis at Week 24 and Week 96
Description: Proportions of subjects in EFX vs placebo groups who achieve resolution of steatohepatitis (defined as a NAS of 0-1 for inflammation, 0 for ballooning, and any value for steatosis) and no worsening of liver fibrosis (determined by the NASH CRN criteria)
Time Frame: 24 and 96 weeks
Population: Liver Biopsy Analysis Set - Week 24 and Week 96
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 41 | 38 | 34
Participants
  Week 24 | 6 | 18 | 26
  Week 96: number analyzed (Participants) | 34 | 26 | 28
  Week 96 | 8 | 16 | 16
Statistical Analysis 1: Comparison: Placebo vs Efruxifermin 28 mg; Week 24; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — Threshold for significance set at p<0.05; A Cochran-Mantel-Haenszel test adjusting for stratification factors was used for comparison between the efruxifermin 28 mg and placebo group; percent difference = 31.9, 95% CI 2-sided [12.9 to 50.9]
Statistical Analysis 2: Comparison: Placebo vs Efruxifermin 50 mg; Week 24; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Threshold for significance set at p<0.05; A Cochran-Mantel-Haenszel test adjusting for stratification factors was used for comparisons between the efruxifermin 50 mg and placebo groups; percent difference = 61.7, 95% CI 2-sided [44.1 to 79.4]
Statistical Analysis 3: Comparison: Placebo vs Efruxifermin 28 mg; Week 96; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — Threshold for significance set at p<0.05; A Cochran-Mantel-Haenszel test adjusting for stratification factors was used for comparisons between efruxifermin 28 mg and placebo groups; percent difference = 38.9, 95% CI 2-sided [17.2 to 60.7]
Statistical Analysis 4: Comparison: Placebo vs Efruxifermin 50 mg; Week 96; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — Threshold for significance set at p<0.05; [statistical method as in outcome 2, analysis 2]; percent difference = 33.2, 95% CI 2-sided [10.5 to 55.8]

4. Secondary Outcome: Proportion of Subjects Who Achieve Improvement in Liver Fibrosis ≥ 1 Stage at Week 24 and Week 96
Description: Proportion of subjects in EFX vs placebo groups who achieve improvement in liver fibrosis (decrease ≥ 1 stage in NASH CRN fibrosis score)
Time Frame: 24 and 96 Weeks
Population: Week 24 and Week 96 Liver Biopsy Analysis Sets
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 41 | 38 | 34
Participants
  Week 24 | 9 | 15 | 14
  Week 96: number analyzed (Participants) | 34 | 26 | 28
  Week 96 | 9 | 12 | 21
Statistical Analysis 1: Comparison: Placebo vs Efruxifermin 28 mg; Week 24; Test type: Superiority; p = 0.053, Cochran-Mantel-Haenszel — Threshold for significance set at p<0.05; [statistical method as in outcome 2, analysis 1]; percent difference = 20.0, 95% CI 2-sided [0.4 to 39.5]
Statistical Analysis 2: Comparison: Placebo vs Efruxifermin 50 mg; Week 24; Test type: Superiority; p = 0.069, Cochran-Mantel-Haenszel — Threshold for statistical significance set at p<0.05; [statistical method as in outcome 3, analysis 2]; percent difference = 19.9, 95% CI 2-sided [-1.5 to 41.2]
Statistical Analysis 3: Comparison: Placebo vs Efruxifermin 28 mg; Week 96; Test type: Superiority; p = 0.123, Cochran-Mantel-Haenszel — Threshold for significance set at p<0.05; A Cochran-Mantel-Haenszel test adjusting for stratification factors was used for comparisons between the efruxifermin 28 mg and placebo groups; percent difference = 19, 95% CI 2-sided [-4.8 to 42.8]
Statistical Analysis 4: Comparison: Placebo vs Efruxifermin 50 mg; Week 96; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Threshold for significance set at p<0.05; [statistical method as in outcome 3, analysis 2]; percent difference = 49.0, 95% CI 2-sided [27.7 to 70.2]

5. Secondary Outcome: Change From Baseline in Hepatic Fat Fraction in EFX vs Placebo Groups
Description: Change from baseline in hepatic fat fraction, measured by magnetic resonance imaging proton-density fat fraction (MRI-PDFF):
  Week 24 and Week 96 MRI-PDFF Analysis Set
Time Frame: 24 and 96 Weeks
Population: Week 24 and 96 MRI-PDFF Analysis Set
Measure: Mean (Standard Error); unit: percentage hepatic fat
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 42 | 38 | 35
percentage hepatic fat
  Week 24 | -1.9 (0.78) | -8.8 (0.84) | -11.2 (0.86)
  Week 96: number analyzed (Participants) | 34 | 26 | 28
  Week 96 | -2.5 (0.89) | -6.3 (1.01) | -8.3 (1.00)
Statistical Analysis 1: Comparison: Placebo vs Efruxifermin 28 mg; Percent change from baseline in hepatic fat fraction between the EFX 28 mg and placebo groups; Test type: Superiority — Week 24; p < 0.001, Mixed Models Analysis — Threshold for significance set at p<0.05; MMRM: fixed effects of treatment, stratification factors, post-baseline visit, treatment-by-visit interaction and baseline as covariate for comparison; Mean Difference (Net) = -6.9, 95% CI 2-sided [-9.09 to -4.71], Standard Error of Mean 1.10
Statistical Analysis 2: Comparison: Placebo vs Efruxifermin 50 mg; Percent change from baseline in hepatic fat fraction between the EFX 50 mg and placebo groups; Test type: Superiority — Week 24; p < 0.001, Mixed Models Analysis — Threshold for significance set at p<0.05; MMRM:fixed effects of treatment, stratification factors, post-baseline visit, treatment-by-visit interaction and baseline as covariates for comparison; Mean Difference (Net) = -9.2, 95% CI 2-sided [-11.47 to -7.02], Standard Error of Mean 1.12
Statistical Analysis 3: Comparison: Placebo vs Efruxifermin 28 mg; Percent change from baseline in hepatic fat fraction between the EFX 28 mg and placebo groups; Test type: Superiority — Week 96; p = 0.005, Mixed Models Analysis — Threshold for significance set at p<0.05; [statistical method as in outcome 5, analysis 2]; Mean Difference (Net) = -3.8, 95% CI 2-sided [-6.39 to -1.18], Standard Error of Mean 1.31
Statistical Analysis 4: Comparison: Placebo vs Efruxifermin 50 mg; Percent change from baseline in hepatic fat fraction between the EFX 50 mg and placebo groups; Test type: Superiority — Week 96; p < 0.001, Mixed Models Analysis — Threshold for significance set at p<0.05; [statistical method as in outcome 5, analysis 2]; Mean Difference (Net) = -5.8, 95% CI 2-sided [-8.38 to -3.25], Standard Error of Mean 1.29

6. Secondary Outcome: Change From Baseline in Lipoproteins at Week 24 and Week 96
Description: Change from baseline of lipoproteins (triglycerides, Non-HDL-C, HDL-C and LDL-C) in EFX vs placebo groups
Time Frame: 24 and 96 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 43 | 42 | 43
mg/dL
  Change from baseline in triglycerides (mg/dL) at Week 24: number analyzed (Participants) | 42 | 35 | 36
  Change from baseline in triglycerides (mg/dL) at Week 24 | 10.5 (6.82) | -41.1 (7.26) | -44.7 (7.20)
  Change from baseline in triglycerides (mg/dL) at Week 96: number analyzed (Participants) | 34 | 26 | 27
  Change from baseline in triglycerides (mg/dL) at Week 96 | 16.1 (7.69) | -26.9 (8.63) | -31.7 (8.54)
  Change from baseline in HDL cholesterol (mg/dL) at Week 24: number analyzed (Participants) | 42 | 35 | 36
  Change from baseline in HDL cholesterol (mg/dL) at Week 24 | -0.9 (1.09) | 10.1 (1.16) | 11.5 (1.15)
  Change from baseline in HDL cholesterol (mg/dL) at Week 96: number analyzed (Participants) | 34 | 26 | 27
  Change from baseline in HDL cholesterol (mg/dL) at Week 96 | 1.3 (1.43) | 7.3 (1.59) | 10.7 (1.57)
  Change from baseline in LDL cholesterol (mg/dL) at Week 24: number analyzed (Participants) | 42 | 35 | 36
  Change from baseline in LDL cholesterol (mg/dL) at Week 24 | 4.0 (3.47) | -10.4 (3.7) | -9.6 (3.69)
  Change from baseline in LDL cholesterol (mg/dL) at Week 96: number analyzed (Participants) | 34 | 26 | 27
  Change from baseline in LDL cholesterol (mg/dL) at Week 96 | -1.3 (4.74) | -1.2 (5.29) | -1.4 (5.23)
  Change from baseline in non-HDL cholesterol (mg/dL) at Week 24: number analyzed (Participants) | 42 | 35 | 36
  Change from baseline in non-HDL cholesterol (mg/dL) at Week 24 | 6.1 (3.83) | -16.6 (4.08) | -16.6 (4.05)
  Change from baseline in non-HDL cholesterol (mg/dL) at Week 96: number analyzed (Participants) | 34 | 26 | 27
  Change from baseline in non-HDL cholesterol (mg/dL) at Week 96 | 1.5 (5.31) | -4.5 (5.92) | -6.7 (5.86)
Statistical Analysis 1: Comparison: Placebo vs Efruxifermin 28 mg; Treatment comparison of least squares (LS) mean change from baseline (EFX 28 mg - placebo) in triglycerides (mg/dL); Test type: Superiority — Week 24; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -51.6, 95% CI 2-sided [-71.17 to -32.11], Standard Error of Mean 9.86
Statistical Analysis 2: Comparison: Placebo vs Efruxifermin 50 mg; Treatment comparison of least squares (LS) mean change from baseline (EFX 50 mg - placebo) in triglycerides (mg/dL); Test type: Superiority — Week 24; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -55.2, 95% CI 2-sided [-74.63 to -35.71], Standard Error of Mean 9.83
Statistical Analysis 3: Comparison: Placebo vs Efruxifermin 28 mg; Treatment comparison of least squares (LS) mean change from baseline (EFX 28 mg - placebo) in triglycerides (mg/dL); Test type: Superiority — Week 96; p < 0.001, Mixed Models Analysis — Threshold for significance set at p<0.05; Mean Difference (Net) = -43.0, 95% CI 2-sided [-65.73 to -20.27], Standard Error of Mean 11.48 — LS Means and differences, SEs, and p-values are from a MMRM with fixed effects of treatment, stratification factors, post-baseline visit, treatment-by-visit interaction, and baseline as a covariate for comparisons between the EFX and placebo group
Statistical Analysis 4: Comparison: Placebo vs Efruxifermin 50 mg; Treatment comparison of LS mean change from baseline (EFX 50 mg - placebo) in triglycerides (mg/dL); Test type: Superiority — Week 96; p < 0.001, Mixed Models Analysis — Threshold for significance set at p<0.05; Mean Difference (Net) = -47.8, 95% CI 2-sided [-70.39 to -25.24], Standard Error of Mean 11.40 — [estimate comment as in outcome 6, analysis 3]
Statistical Analysis 5: Comparison: Placebo vs Efruxifermin 28 mg; Treatment comparison of LS mean change from baseline (EFX 28 mg - placebo) in HDL cholesterol (mg/dL); Test type: Superiority — Week 24; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 11.0, 95% CI 2-sided [7.92 to 14.17], Standard Error of Mean 1.58
Statistical Analysis 6: Comparison: Placebo vs Efruxifermin 50 mg; Treatment comparison of LS mean change from baseline (EFX 50 mg - placebo) in HDL cholesterol (mg/dL); Test type: Superiority — Week 24; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 12.5, 95% CI 2-sided [9.35 to 15.57], Standard Error of Mean 1.57
Statistical Analysis 7: Comparison: Placebo vs Efruxifermin 28 mg; Treatment comparison of LS mean change from baseline (EFX 28 mg - placebo) in HDL cholesterol (mg/dL); Test type: Superiority — Week 96; p = 0.005, Mixed Models Analysis — Threshold for significance set at p<0.05; Mean Difference (Net) = 6.0, 95% CI 2-sided [1.84 to 10.23], Standard Error of Mean 2.12 — [estimate comment as in outcome 6, analysis 3]
Statistical Analysis 8: Comparison: Placebo vs Efruxifermin 50 mg; Treatment comparison of LS mean change from baseline (EFX 50 mg - placebo) in HDL cholesterol (mg/dL); Test type: Superiority — Week 96; p < 0.001, Mixed Models Analysis — Threshold for significance set at p<0.05; Mean Difference (Net) = 9.5, 95% CI 2-sided [5.30 to 13.65], Standard Error of Mean 2.11 — [estimate comment as in outcome 6, analysis 3]
Statistical Analysis 9: Comparison: Placebo vs Efruxifermin 28 mg; Treatment comparison of change from baseline (EFX 28 mg - placebo) in LDL cholesterol (mg/dL); Test type: Superiority — Week 24; p = 0.005, Mixed Models Analysis; Mean Difference (Net) = -14.4, 95% CI 2-sided [-24.28 to -4.53], Standard Error of Mean 4.99
Statistical Analysis 10: Comparison: Placebo vs Efruxifermin 50 mg; Treatment comparison of LS mean change from baseline (EFX 50 mg - placebo) in LDL cholesterol (mg/dL); Test type: Superiority — Week 24; p = 0.007, Mixed Models Analysis; Median Difference (Net) = -13.6, 95% CI 2-sided [-23.50 to -3.76], Standard Error of Mean 4.98
Statistical Analysis 11: Comparison: Placebo vs Efruxifermin 28 mg; Treatment comparison of change from baseline (EFX 28 mg - placebo) in LDL cholesterol (mg/dL); Test type: Superiority — Week 96; p = 0.990, Mixed Models Analysis — Threshold for significance set at p<0.05; Mean Difference (Net) = 0.1, 95% CI 2-sided [-13.86 to 14.04], Standard Error of Mean 7.04 — [estimate comment as in outcome 6, analysis 3]
Statistical Analysis 12: Comparison: Placebo vs Efruxifermin 50 mg; Treatment comparison of LS mean change from baseline (EFX 50 mg - placebo) in LDL cholesterol (mg/dL); Test type: Superiority — Week 96; p = 0.980, Mixed Models Analysis — Threshold for significance set at p<0.05; Mean Difference (Net) = -0.2, 95% CI 2-sided [-14.07 to 13.71], Standard Error of Mean 7.01 — [estimate comment as in outcome 6, analysis 3]
Statistical Analysis 13: Comparison: Placebo vs Efruxifermin 28 mg; Treatment comparison of LS mean change from baseline (EFX 28 mg - placebo) in non-HDL cholesterol (mg/dL); Test type: Superiority — Week 24; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -22.6, 95% CI 2-sided [-33.58 to -11.71], Standard Error of Mean 5.52
Statistical Analysis 14: Comparison: Placebo vs Efruxifermin 50 mg; Treatment comparison of LS mean change from baseline (EFX 50mg - placebo) in non-HDL cholesterol (mg/dL); Test type: Superiority — Week 24; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -22.7, 95% CI 2-sided [-33.56 to -11.74], Standard Error of Mean 5.51
Statistical Analysis 15: Comparison: Placebo vs Efruxifermin 28 mg; Treatment comparison of LS mean change from baseline (EFX 28 mg - placebo) in non-HDL cholesterol (mg/dL); Test type: Superiority — Week 96; p = 0.443, Mixed Models Analysis — Threshold for significance set at p<0.05; Mean Difference (Net) = -6.1, 95% CI 2-sided [-21.72 to 9.56], Standard Error of Mean 7.90 — [estimate comment as in outcome 6, analysis 3]
Statistical Analysis 16: Comparison: Placebo vs Efruxifermin 50 mg; Treatment comparison of LS mean change from baseline (EFX 50 mg - placebo) in non-HDL cholesterol (mg/dL); Test type: Superiority — Week 96; p = 0.299, Mixed Models Analysis — Threshold for significance set at p<0.05; Mean Difference (Net) = -8.2, 95% CI 2-sided [-23.77 to 7.36], Standard Error of Mean 7.86 — [estimate comment as in outcome 6, analysis 3]

7. Secondary Outcome: Change From Baseline of Hemoglobin A1c (Glycated Hemoglobin, HbA1c) at Week 24 and Week 96
Description: Change from baseline in hemoglobin A1c (glycated hemoglobin, HbA1c) in EFX vs placebo groups
Time Frame: 24 Weeks, 96 Weeks
Population: Biomarker Analysis Set
Measure: Least Squares Mean (Standard Error); unit: % glycated hemoglobin
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 43 | 40 | 43
% glycated hemoglobin
  Change from baseline in hemoglobin A1C (HbA1c, %) at Week 24: number analyzed (Participants) | 42 | 37 | 36
  Change from baseline in hemoglobin A1C (HbA1c, %) at Week 24 | -0.0 (0.12) | -0.3 (0.12) | -0.4 (0.12)
  Change from baseline in hemoglobin A1C (HbA1c, %) at Week 96: number analyzed (Participants) | 34 | 27 | 27
  Change from baseline in hemoglobin A1C (HbA1c, %) at Week 96 | -0.0 (0.22) | 0.0 (0.24) | 0.2 (0.24)

8. Secondary Outcome: Change From Baseline in C-peptide at Week 24 and Week 96
Description: Change from baseline in C-peptide in EFX vs placebo groups
Time Frame: 24 Weeks, 96 Weeks
Population: Biomarker Analysis Set
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 43 | 40 | 43
ng/mL
  Change from baseline in C-Peptide at Week 24: number analyzed (Participants) | 41 | 37 | 36
  Change from baseline in C-Peptide at Week 24 | 0.0 (0.19) | -0.8 (0.20) | -1.2 (0.19)
  Change from baseline in C-Peptide at Week 96: number analyzed (Participants) | 35 | 28 | 27
  Change from baseline in C-Peptide at Week 96 | -0.2 (0.22) | -0.4 (0.25) | -1.0 (0.25)

9. Secondary Outcome: Change From Baseline in Adiponectin at Week 24 and Week 96
Description: Change from baseline in adiponectin in EFX vs placebo groups
Time Frame: 24 Weeks, 96 Weeks
Population: Biomarker Analysis Set
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 43 | 40 | 43
ng/mL
  Change from baseline in adiponectin at Week 24: number analyzed (Participants) | 42 | 36 | 34
  Change from baseline in adiponectin at Week 24 | 296.4 (312.56) | 1411.5 (333.48) | 3088.8 (333.82)
  Change from baseline in adiponectin at Week 96: number analyzed (Participants) | 35 | 27 | 27
  Change from baseline in adiponectin at Week 96 | 531.5 (416.93) | 975.3 (459.40) | 2018.3 (458.91)

10. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at Week 24 and Week 96
Description: Change from baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) in EFX vs placebo groups
  The Homeostatic Model Assessment of Insulin Resistance, HOMA-IR, is a calculated index that estimates insulin resistance based on fasting glucose and insulin levels. Higher values indicate greater insulin resistance.
  < 1.0: Normal insulin sensitivity 1.0-1.9: Mild insulin resistance 2.0-2.9: Moderate insulin resistance > 2.9: Severe insulin resistance
Time Frame: 24 Weeks, 96 Weeks
Population: Biomarker Analysis Set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 43 | 40 | 43
units on a scale
  Change from baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at Week 24: number analyzed (Participants) | 39 | 32 | 34
  Change from baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at Week 24 | 0.7 (1.09) | -4.7 (1.19) | -5.6 (1.14)
  Change from baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at Week 96: number analyzed (Participants) | 34 | 25 | 26
  Change from baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at Week 96 | -1.3 (0.87) | -4.1 (1.01) | -5.5 (0.99)

11. Secondary Outcome: Change From Baseline in Enhanced Liver Fibrosis (ELF) Score at Week 24 and Week 96
Description: Change from Baseline in Enhanced Liver Fibrosis (ELF) Score in EFX vs placebo groups
  The Enhanced Liver Fibrosis (ELF) score is a non-invasive blood test that assesses the risk of liver fibrosis and its progression.
  Lower risk (<9.8): Suggests a lower risk of advanced liver fibrosis. Mid risk (9.8-11.2): Indicates a moderate risk of disease progression. Higher risk (≥11.3): Suggests a higher risk of developing cirrhosis or liver-related events
Time Frame: 24 and 96 Weeks
Population: Biomarker Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 43 | 40 | 43
score on a scale
  Change from baseline in ELF Score at Week 24: number analyzed (Participants) | 42 | 37 | 34
  Change from baseline in ELF Score at Week 24 | 0.1 (0.10) | -0.6 (0.10) | -0.7 (0.10)
  Change from baseline in ELF Score at Week 96: number analyzed (Participants) | 35 | 27 | 25
  Change from baseline in ELF Score at Week 96 | -0.1 (0.14) | -0.7 (0.16) | -0.8 (0.16)

12. Secondary Outcome: Change From Baseline in N-terminal Type III Collagen Propeptide (Pro-C3) at Week 24 and Week 96
Description: Change from Baseline in N-terminal Type III Collagen Propeptide (Pro-C3) in EFX vs placebo groups
Time Frame: 24 and 96 Weeks
Population: Biomarker Analysis Set
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 43 | 40 | 43
ng/mL
  Change from baseline in N-terminal Type III Collagen Propeptide (Pro-C3) GEN2 at Week 24: number analyzed (Participants) | 42 | 37 | 36
  Change from baseline in N-terminal Type III Collagen Propeptide (Pro-C3) GEN2 at Week 24 | -2.7 (6.99) | -51.1 (7.37) | -53.9 (7.37)
  Change from baseline in N-terminal Type III Collagen Propeptide (Pro-C3) GEN2 at Week 96: number analyzed (Participants) | 35 | 27 | 27
  Change from baseline in N-terminal Type III Collagen Propeptide (Pro-C3) GEN2 at Week 96 | -17.2 (7.87) | -40.2 (8.89) | -50.5 (8.92)

13. Secondary Outcome: Change From Baseline in Collagen III Neo-Peptide (C3M) at Week 24 and Week 96
Description: Change from Baseline in Collagen III Neo-Peptide (C3M) in EFX vs placebo groups
Time Frame: 24 and 96 Weeks
Population: Biomarker Analysis Set
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 43 | 40 | 43
ng/mL
  Change from baseline in Collagen III Neo-Peptide (C3M) (ng/mL) at Week 24: number analyzed (Participants) | 42 | 37 | 36
  Change from baseline in Collagen III Neo-Peptide (C3M) (ng/mL) at Week 24 | 0.2 (0.35) | -0.8 (0.37) | -1.1 (0.38)
  Change from baseline in Collagen III Neo-Peptide (C3M) (ng/mL) at Week 96: number analyzed (Participants) | 35 | 27 | 27
  Change from baseline in Collagen III Neo-Peptide (C3M) (ng/mL) at Week 96 | 3.1 (0.71) | 3.3 (0.80) | 4.4 (0.80)

14. Secondary Outcome: Change From Baseline in NIS4 Score at Week 24 and Week 96
Description: Change from Baseline in NIS4 score in EFX vs placebo groups
  NIS4 scores range from 0 to 1 and are calculated by combining the results of four individual biomarker assays [miR34a-5p, α2-macroglobulin (A2M), YKL-40 and HbA1c] each of which contributes to the test's ability to detect liver inflammation and/or fibrosis.
  >0.63: Higher risk of NASH or advanced fibrosis 0.37-0.63: Moderate risk, and additional testing may be considered <0.36: Lower risk of of NASH or advanced fibrosis
Time Frame: 24 and 96 Weeks
Population: Biomarker Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 43 | 40 | 43
score on a scale
  Change from baseline in NIS-4 score at Week 24: number analyzed (Participants) | 39 | 35 | 31
  Change from baseline in NIS-4 score at Week 24 | -0.0 (0.03) | -0.3 (0.04) | -0.3 (0.04)
  Change from baseline in NIS-4 score at Week 96: number analyzed (Participants) | 31 | 26 | 24
  Change from baseline in NIS-4 score at Week 96 | -0.1 (0.05) | -0.2 (0.05) | -0.3 (0.05)

15. Secondary Outcome: Change in Body Weight at Week 24 and Week 96
Description: Change from baseline in body weight (kg) in EFX vs placebo groups
Time Frame: 24 and 96 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 43 | 42 | 43
kg
  Change from Baseline in Body Weight (kg) at Week 24: number analyzed (Participants) | 42 | 37 | 36
  Change from Baseline in Body Weight (kg) at Week 24 | -0.6 (0.82) | -0.2 (0.86) | -3.0 (0.85)
  Change from Baseline in Body Weight (kg) at Week 96: number analyzed (Participants) | 34 | 27 | 27
  Change from Baseline in Body Weight (kg) at Week 96 | -1.5 (1.40) | -0.3 (1.53) | -3.5 (1.52)
Statistical Analysis 1: Comparison: Placebo vs Efruxifermin 28 mg; Treatment comparison of LS mean change from baseline (EFX 28 mg - placebo) in body weight (kg); Test type: Superiority — Week 24; p = 0.750, Mixed Models Analysis — Threshold for significance set at p<0.05; Mean Difference (Net) = 0.4, 95% CI 2-sided [-1.96 to 2.72], Standard Error of Mean 1.18
Statistical Analysis 2: Comparison: Placebo vs Efruxifermin 50 mg; Treatment comparison of LS mean change from baseline (EFX 50 mg - placebo) in body weight (kg); Test type: Superiority — Week 24; p = 0.042, Mixed Models Analysis — Threshold for significance set at p<0.05; Mean Difference (Net) = -2.4, 95% CI 2-sided [-4.75 to -0.09], Standard Error of Mean 1.18
Statistical Analysis 3: Comparison: Placebo vs Efruxifermin 28 mg; Treatment comparison of LS mean change from baseline (28 mg EFX - placebo) in body weight (kg); Test type: Superiority — Week 96; p = 0.564, Mixed Models Analysis; Mean Difference (Net) = 1.2, 95% CI 2-sided [-2.90 to 5.29], Standard Error of Mean 2.07
Statistical Analysis 4: Comparison: Placebo vs Efruxifermin 50 mg; Treatment comparison of LS mean change from baseline (EFX 50 mg - placebo) in body weight (kg); Test type: Superiority — Week 96; p = 0.348, Mixed Models Analysis; Mean Difference (Net) = -1.9, 95% CI 2-sided [-6.02 to 2.14], Standard Error of Mean 2.06

16. Secondary Outcome: Change From Baseline in Liver Stiffness (kPa) at Week 24 and Week 96
Description: Change from Baseline in Liver Stiffness Evaluated by FibroScan in EFX vs placebo groups at Week 24 and Week 96:
  Full Analysis Set
Time Frame: 24 and 96 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: kPa
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
Number analyzed (Participants) | 43 | 42 | 43
kPa
  Change from baseline in liver stiffness measurement (LSM, kPa) at Week 24: number analyzed (Participants) | 42 | 38 | 37
  Change from baseline in liver stiffness measurement (LSM, kPa) at Week 24 | -0.8 (0.88) | -2.9 (0.93) | -4.2 (0.95)
  Change from baseline in liver stiffness measurement (LSM, kPa) at Week 96: number analyzed (Participants) | 33 | 27 | 28
  Change from baseline in liver stiffness measurement (LSM, kPa) at Week 96 | -0.6 (0.98) | -4.0 (1.09) | -7.2 (1.08)
Statistical Analysis 1: Comparison: Placebo vs Efruxifermin 28 mg; Treatment comparison of change from baseline (EFX 28 mg - placebo) in Liver Stiffness Measurement (kPa); Test type: Superiority — Week 24; p = 0.102, Mixed Models Analysis; Mean Difference (Net) = -2.1, 95% CI 2-sided [-4.5 to 0.4], Standard Error of Mean 1.24
Statistical Analysis 2: Comparison: Placebo vs Efruxifermin 50 mg; Treatment comparison of change from baseline (EFX 50 mg - placebo) in Liver Stiffness Measurement (kPa); Test type: Superiority — Week 24; p = 0.009, Mixed Models Analysis; Mean Difference (Net) = -3.3, 95% CI 2-sided [-5.8 to -0.8], Standard Error of Mean 1.26
Statistical Analysis 3: Comparison: Placebo vs Efruxifermin 28 mg; Treatment comparison of change from baseline (EFX 28 mg - placebo) in Liver Stiffness Measurement (kPa); Test type: Superiority — Week 96; p = 0.021, Mixed Models Analysis — Threshold for significance set at P<0.05; Mean Difference (Net) = -3.4, 95% CI 2-sided [-6.2 to -0.5], Standard Error of Mean 1.43 — LS Means, SEs, and p-values are from a MMRM with fixed effects of treatment, stratification factors, post-baseline visit, treatment-by-visit interaction, and baseline as a covariate for comparisons between the EFX 28 mg and placebo group
Statistical Analysis 4: Comparison: Placebo vs Efruxifermin 50 mg; Treatment comparison of change from baseline (EFX 50 mg - placebo) in Liver Stiffness Measurement (kPa); Test type: Superiority — Week 96; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -6.6, 95% CI 2-sided [-9.4 to -3.7], Standard Error of Mean 1.43 — LS Means, SEs, and p-values are from a MMRM with fixed effects of treatment, stratification factors, post-baseline visit, treatment-by-visit interaction, and baseline as a covariate for comparisons between the EFX 50 mg and placebo group

ADVERSE EVENTS:
Time Frame: 96 weeks
Arm/Group | Placebo | Efruxifermin 28 mg | Efruxifermin 50 mg
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/40 | 0/43
Serious Adverse Events (participants affected / at risk) | 4/43 | 4/40 | 7/43
Other Adverse Events (participants affected / at risk) | 42/43 | 38/40 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | Efruxifermin 28 mg (N=40) | Efruxifermin 50 mg (N=43)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Esophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis, necrotizing (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Face edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | Efruxifermin 28 mg (N=40) | Efruxifermin 50 mg (N=43)
Diarrhea (Gastrointestinal disorders) | 13 | 23 | 19
Nausea (Gastrointestinal disorders) | 13 | 16 | 19
COVID-19 (Infections and infestations) | 13 | 10 | 16
injection-site erythema (General disorders) | 8 | 10 | 8
Vomiting (Gastrointestinal disorders) | 7 | 8 | 8
Increased appetite (Metabolism and nutrition disorders) | 3 | 8 | 10
Injection-site bruising (General disorders) | 7 | 8 | 6
Procedural pain (Injury, poisoning and procedural complications) | 7 | 8 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 7 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 6
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 7
Headache (Nervous system disorders) | 6 | 6 | 5
Type 2 diabetes (Metabolism and nutrition disorders) | 8 | 4 | 4
Sinusitis (Infections and infestations) | 7 | 3 | 5
Hypertension (Vascular disorders) | 1 | 8 | 5
Nasopharyngitis (Infections and infestations) | 6 | 6 | 1
Abdominal pain, upper (Gastrointestinal disorders) | 5 | 2 | 4
Constipation (Gastrointestinal disorders) | 3 | 5 | 3
Abdominal distension (Gastrointestinal disorders) | 3 | 3 | 4
Frequent bowel movements (Gastrointestinal disorders) | 1 | 9 | 0
Flatulence (Gastrointestinal disorders) | 3 | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 5 | 2
Toothache (Gastrointestinal disorders) | 1 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 4 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 3 | 0
Influenza (Infections and infestations) | 5 | 1 | 2
Urinary tract infection (Infections and infestations) | 2 | 4 | 1
Fatigue (General disorders) | 5 | 4 | 3
Injection site pruritus (General disorders) | 2 | 4 | 6
Injection-site reaction (General disorders) | 3 | 5 | 3
Injection-site rash (General disorders) | 1 | 3 | 6
Early satiety (General disorders) | 3 | 3 | 1
Swelling face (General disorders) | 0 | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 5 | 2 | 4
Fall (Injury, poisoning and procedural complications) | 5 | 2 | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 3 | 2
Dizziness (Nervous system disorders) | 4 | 2 | 2
Migraine (Nervous system disorders) | 3 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 3
Depression (Psychiatric disorders) | 2 | 2 | 4
Anxiety (Psychiatric disorders) | 0 | 5 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 3 | 2
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication of the Study results by Sponsor, or if a publication is not submitted within 18 months after conclusion, the Investigator may publish or present the results of Institution's and Investigator's activities conducted under this Agreement. Investigator agrees to submit any proposed publication or presentation to Sponsor for review at least 90 days prior to submitting.

DOCUMENTS (2):
  • Study Protocol (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT04767529/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT04767529/SAP_001.pdf